CLINICAL TRIAL: NCT05085574
Title: A Phase 2 Randomized, Single-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of the Combination of Famotidine and Celecoxib as a Treatment in Moderate-to-severe Patients Hospitalized for COVID-19
Brief Title: Leidos-Enabled Adaptive Protocol for Clinical Trials (LEAP-CT) in Hospitalized Patients With COVID-19 (Addendum 1)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID environment, lack of site confidence to enroll subjects, sites not suited to study procedures, decline of potential inpatient subjects at site
Sponsor: Leidos Life Sciences (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LDOS-21-001-01
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: 2019 Novel Coronavirus Disease; 2019 Novel Coronavirus Infection; 2019-nCoV Disease; 2019-nCoV Infection; COVID-19 Pandemic; COVID-19 Virus Disease; COVID-19 Virus Infection; Covid19; Coronavirus Disease 2019; SARS-CoV-2 Infection; SARS-CoV-2 Acute Respiratory Disease; COVID-19
Keywords: COVID-19; COVID; COVID19; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Famotidine; Celecoxib

STUDY DESIGN:
Intervention Model Description: Subjects randomized 1:1, study drug:placebo
Who Masked: Participant
Masking Description: Single-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Study Product) (Experimental): Subjects will receive 80 mg famotidine (PO) QID and 400 mg celecoxib as a first dose, followed by 200 mg (PO) BID celecoxib, for 5 days. Following this 5-day period, subjects will continue their famotidine treatment for an additional 9 days.
  Interventions: Drug: Famotidine; Drug: Celecoxib
- Group 2 (Reference Therapy) (Placebo Comparator): Subjects will receive matching placebos QID and BID, for 5 days. Following this 5-day period, subjects will continue to receive matching famotidine placebo, QID, for an additional 9 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Famotidine — 80 mg tablet, QID for 14 days
  Other Names: Pepcid
  Arms: Group 1 (Study Product)
Drug: Celecoxib — 400 mg (initial dose), then 200 mg capsule, BID for 5 days
  Other Names: Celebrex
  Arms: Group 1 (Study Product)
Drug: Placebo — tablet, QID for 14 days; capsule, BID for 5 days
  Arms: Group 2 (Reference Therapy)

SUMMARY:
This study is designed to test the efficacy and safety of combinations of two well-understood agents - famotidine and celecoxib in patients hospitalized with moderate-to-severe COVID-19 (based on World Health Organization [WHO] Ordinal Scale for Clinical Improvement). Both famotidine and celecoxib separately demonstrate clinical activity in mitigating COVID-19 disease symptoms or severity, and appear to have separate and complementary mechanisms of action.

DETAILED DESCRIPTION:
Participants will be randomly assigned, in a 1:1 ratio, to one of two regimens, with 202 subjects per group as follows:

Group 1 (study product) subjects will receive 80 mg famotidine by mouth (PO) 4 times per day (QID) + 400 mg celecoxib as a first dose, followed by 200 mg celecoxib PO, 2 times per day (BID), for 5 days. Following this 5-day period, subjects will continue their famotidine treatment for an additional 9 days.

Group 2 (reference therapy) subjects will receive matching placebos QID and BID, for 5 days. Following this 5-day period, subjects will continue to receive matching famotidine placebo, QID, for an additional 9 days.

Safety, efficacy and pharmacokinetics of famotidine and celecoxib will be evaluated.

All participants will receive the standard of care (SOC), which typically consists of remdesivir, decadron (dexamethasone), lovenox, tociluzimab, and convalescent plasma. At the discretion of the investigator, study treatment can be stopped and dexamethasone initiated in study participants who require supplemental oxygen (WHO 5) as outlined in the NIH COVID-19 Treatment Guidelines. Investigators are required to stop study treatment and initiate dexamethasone, as indicated in participants who require high-flow oxygen (WHO 6), non-invasive ventilation (NIV; WHO 6), invasive mechanical ventilation (WHO 7-8) or extracorporeal membrane oxygenation (ECMO; WHO 9), in accordance with the NIH COVID-19 Treatment Guidelines. The NIH COVID-19 Treatment Guidelines recommend against the use of dexamethasone only in hospitalized patients not requiring supplemental oxygen (WHO 4).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants must be at least 18 years of age, inclusive, at the time of signing the informed consent form.
* Confirmed COVID-19 or symptom onset within 7 days of hospitalization, as shown by medical history, physical exam, and laboratory tests (PCR), and who have been hospitalized for COVID-19 at WHO Grade 4-5.
* Contraceptive use by men or women should be consistent with Appendix 4 of the Master Protocol (LDOS-21-001).
* Capable of understanding and providing a signed informed consent form.
* Reliable access to the internet.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Pregnant or breastfeeding
* History of HIV
* Ongoing treatment that cannot be temporarily discontinued during the study: anti-inflammatory treatment (nonsteroidal anti-inflammatory drugs [NSAIDS]);corticosteroids; antimalarials; antiarrhythmics; tricyclic antidepressants; natalizumab; quinolones; macrolides; and agalsidase alfa and beta

  1. drugs dependent on gastric pH for absorption, e.g., dasatinib, delavirdine, mesylate, cefditoren, and fosamprenavir;
  2. tizanidine (CYP1A2) substrate;
  3. drugs that interfere with hemostasis (e.g., warfarin, aspirin, selective serotonin reuptake inhibitors [SSRIs]/serotonin norepinephrine reuptake inhibitors [SNRIs]);
  4. angiotensin converting enzyme (ACE) inhibitors, angiotensin receptor blockers (ARB), or beta-blockers;
  5. diuretics;
  6. digoxin
* Ongoing famotidine, celecoxib, or other COVID-19 clinical investigational treatment(s) within the past 30 days or current participation in another investigational clinical trial
* History of immunosuppression
* History of asthma, urticaria, or other allergic-type reactions after taking aspirin or other NSAIDs
* Rejection of participation at the discretion of the Principal Investigator or Sponsor
* Any contraindication for famotidine or celecoxib treatment:

  a. Famotidine or celecoxib hypersensitivity; b. Retinopathy, visual field or visual acuity disturbances; c. History of cardiovascular disease, such as congestive heart failure, QT prolongation, bradycardia (<50 bpm), ventricular tachycardia, other arrhythmias, as determined at screening electrocardiogram (ECG) or medical history; d. Potassium <3 mEq/L (milliequivalent/liter) as determined at Visit 1; e. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >5 upper normal limit, as determined at Visit 1; f. Previous myocardial infarction; e. Myasthenia gravis; h. Psoriasis or porphyria; i. Glomerular clearance, 60 mL/min; j. Previous history of severe hypoglycemia; k. Known or suspected to be poor CYP2C9 metabolizers based on genotype or previous history or experience with other CYP2C9 substrates, such as warfarin and phenytoin; l. Moderate or severe hepatic impairment, e.g., Child-Pugh Class B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Time-to-event to achieve WHO level ≤3 | 30 days
  Evaluation of the time-to-event to achieve a WHO level score ≤3
Death rate | 30 days
  Evaluation of the time-to-event where all-cause mortality occurs

SECONDARY OUTCOMES:
Hospital discharge to chronic palliative care | 30 days
  Measured incidence of hospital discharge to chronic palliative care
Hospital discharge with no additional medical care | 30 days
  Measured incidence of hospital discharge with no additional medical care required
Related adverse events (AEs) and serious adverse events (SAEs) | 90 days
  Measured incidence of related AEs and SAEs
Study discontinuation due to related AEs or SAEs | 90 days
  Measured incidence of study discontinuation due to related AEs or SAEs

OTHER OUTCOMES:
Pharmacokinetic (PK) endpoint-Assess area under the curve | 14 days
  Measure area under the curve (AUC) for famotidine and celecoxib combination in 10 patients per group
Pharmacokinetic (PK) endpoint-Assess time to maximum plasma concentration | 14 days
  Measure time to maximum plasma concentration (tmax) for famotidine and celecoxib combination in 10 patients per group
Pharmacokinetic (PK) endpoint-Assess maximum serum concentration | 14 days
  Measure maximum serum concentration (Cmax) for famotidine and celecoxib combination in 10 patients per group
Exploratory endpoint-Incidence of symptom reduction | 14 days
  Cumulative incidence of clinically significant symptom reduction (severity and duration) using COVID-19 Symptom Score
Exploratory endpoint-Incidence of clinical improvement | 14 days
  Cumulative incidence of clinically significant symptom reduction (severity and duration) using WHO Ordinal Scale for Clinical Improvement
Special Assessment - High-resolution computed tomography (HRCT), 20 patients/group, change from baseline | Study Day 1 (baseline), Day 16 (discharge), 30 days after first dose, and 90 days after first dose
  HRCT scan of the chest
Special Assessment - Total lung capacity (TLC), 20 patients/group, change from baseline | Study Day 1 (baseline), 16 (discharge), 30 days after first dose, and 90 days after first dose
  TLC
Special Assessment - Prostaglandin E2 (PGE2), 20 patients/group, change from baseline | Study Day 1 (baseline), 16 (discharge), 30 days after first dose, and 90 days after first dose
  PGE2 testing
Special Assessments - Urinalysis, 20 patients/group, change from baseline | Study Day 1 (baseline) and 16 (discharge)
  Urinalysis

CONTACTS AND LOCATIONS:
Overall Officials: Tilly Lawrence, BSN, RN, Study Director — Leidos, Inc.

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make individual participant data (IPD) available.